CLINICAL TRIAL: NCT03494244
Title: Post-operative Outcomes as Clinical Evidence for Soft Tissue Reinforcement: a Prospective Cohort Study.
Brief Title: Evaluation of ADM Soft Tissue Reinforcement
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Chienwei Eric Liao, Associate Professor or Surgery, Division of Plastic and Reconstructive Surgery, Massachusetts General Hospital
Other Study IDs: 2018P000084
Record Dates: First submitted 2018-03-08; First posted 2018-04-11 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Breast Cancer; Surgery; Surgical Item, Retained
Keywords: acellular dermal matrix; breast reconstruction; efficacy
MeSH Terms: conditions — Breast Neoplasms; Foreign Bodies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- ADM: Patients having undergone direct-to-implant breast reconstruction using acellular dermal matrix.
  Interventions: Procedure: Direct-to-implant breast reconstruction; Device: Acellular dermal matrix
- Non-ADM (Vicryl): Patients having undergone direct-to-implant breast reconstruction using non-acellular dermal matrix mesh (Vicryl mesh).
  Interventions: Procedure: Direct-to-implant breast reconstruction

INTERVENTIONS:
Procedure: Direct-to-implant breast reconstruction — Terminal prosthetic implanted at the time of mastectomy.
  Other Names: DTI
Device: Acellular dermal matrix — Banked tissue used to support the directly implanted breast prosthesis.
  Other Names: ADM
  Groups: ADM

SUMMARY:
The use of acellular dermal matrix (ADM) has facilitated implant-based breast reconstruction, both in single-stage direct-to-implant (DTI) and staged tissue expander placement. Nearly half of all breast reconstruction procedures performed within the United States have incorporated ADM. Despite such widespread acceptance among both patients and plastic surgeons, manufacturers of ADM face difficulties in obtaining approval by the Food and Drug Administration (FDA) for use of their product as a medical device in breast reconstructions. ADM is defined as banked tissue and, as such, is approved for use as tissue support. Under section 510k of the Food, Drug and Cosmetic Act, ADM must exhibit "soft tissue reinforcement of integument" to be considered a medical device, a criterion that has yet to be physiologically or clinically defined. This distinction precludes the development and manufacture of xenogeneic ADM. The aim of this research is to compare reconstruction outcomes between ADM and Vicryl, a non-ADM control that is hydrolyzed and degraded within 6-8 weeks after surgery. The investigators propose a prospective cohort study to determine whether post-operative outcomes provide clinical and anatomic evidence for soft tissue reinforcement within the ADM group.

DETAILED DESCRIPTION:
This study will measure objective clinical endpoints in DTI breast reconstruction. A total of 152 patients (76 for both ADM and non-ADM cohorts) will be followed in a prospectively recorded database. The clinical care of the patient will be safe-guarded to proceed entirely unaffected by the study. Enrollment will be limited to patients of Dr. Liao and Dr. William Austen at the Massachusetts General Hospital who are scheduled to undergo immediate, DTI breast reconstruction. Patients may undergo immediate, DTI breast reconstruction if they have mastectomies for the purpose of either removing breast cancer or prophylactic removal of the breasts following diagnosis of genetic predisposition for breast cancer based on family history or genetic testing. All patients will be women. The age minimum is 18 years. There is no age maximum.

The study will involve only recording of data (patient characteristics, clinical data, reconstructive parameters (size of ADM and implant used), drain placement, number and caliber of drains, outcomes of surgery). At initial consultation, per the standard routine for Dr. Liao's patients, digital photographs and 3D photographs will be obtained below the neck, eliminating any patient identifiers. Patients will be followed per routine care protocol. A typical patient will be followed weekly for 6 weeks, then at 3 months, 6 months, and 12 months. All photographs are de-identified and taken below the neck, and are kept in a secure photograph database maintained by the Division of Plastic and Reconstructive Surgery. The clinical care of the patient adheres strictly to the existing standard of care by the surgeon (Dr. Liao). The study will involve only the recording of data without any additional interaction with the patient.

The primary clinical endpoint to be measured is breast form. Secondary clinical endpoints include: seroma, infection, skin necrosis, wound problems, explantation, and any other minor or major complications. Breast thickness and landmark positioning will be recorded as quantitative measures of breast form. The investigators will determine tissue thickness in the following areas: (a) point of maximal projection, (b) inferior pole of the breast, and (c) the midpoint between the aforementioned areas, a and b. Measurements will be made using transcutaneous ultrasound (GE NextGen LOGIQ e R7 compact digital ultrasound). Landmark mapping will be conducted via Vectra imaging software. The positioning of the nipples and inframammary fold (IMF) relative to the sternal notch will be determined through a predetermined Vectra algorithm. Post-operative imaging will be conducted at 6 weeks, 3 months, 6 months, and 12 months. Digital images will provide objective information on aesthetic outcomes and evidence of ptosis, pseudoptosis, symmetry, chest position, or nipple position (if nipple sparing) for both cohorts.

In addition to objective clinical outcomes, patient reported outcomes (PRO) will be measured with the Breast-Q questionnaire. The survey will be administered during the initial consult (pre-mastectomy module) and then reassessed (post-mastectomy module) at 3 months (early recovery) and 12 months (late recovery) to track changes in quality of life (QOL). The PRO will be compared between the ADM and non-ADM cohorts.

The investigators expect to reach the goal of 152 patients within 6 to 12 months, and complete the study with a minimum of 6 months of follow-up within 24 months.

ELIGIBILITY:
Inclusion Criteria:

* direct to implant breast reconstruction

Exclusion Criteria:

* BMI > 30
* history of smoking within 1 year of enrollment
* previous breast surgery
* malnutrition or cachexia
* breast implant volume ≤ 125 mL or ≥ 700 mL

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female.
Study Population: patients who undergo breast reconstruction if they have mastectomies for the purpose of either removing breast cancer or prophylactic removal of the breasts following diagnosis of genetic predisposition for breast cancer based on family history or genetic testing
Sampling Method: Non-Probability Sample
Enrollment: 152 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in Tissue thickness (measured in millimeters). | Post-surgical, follow-up intervals extending to one year following reconstruction. Measurements will be performed at the following intervals, post-operatively: 6 weeks, 3 months, 6 months, 12 months.
  Anatomic measurement of mastectomy skin flap thickness will be conducted comparing ADM and Vicryl patient cohorts. Breast skin flap thickness will be measured at landmarks reproducible over time and comparable between patients. We will determine tissue thickness in the following areas: (a) point of maximal projection, (b) the midpoint between maximal projection and the inferior pole of the breast, and (c) the inferior pole of the breast. During measurement, patients will be positioned upright, such that gravitational force will be exerted on the breast skin flap by the prosthesis. Tissue thickness will be determined via transcutaneous ultrasound (GE NextGen LOGIQ e R7 compact digital ultrasound). The mastectomy skin flap will be defined as the tissue between the air-skin interface to the deep margin of the subcutaneous layer. Tissue thickness, in millimeters (mm), will be calculated using a predetermined prediction algorithm.
Change in Anatomic landmark position (measured in centimeters) | Post-surgical, follow-up intervals extending to one year following reconstruction. These cardinal landmarks of breast form and axis length will be collected at the following intervals, post-operatively: 6 weeks, 3 months, 6 months, 12 months.
  Thoracoabdominal images will be captured using Vectra 3M, a three-dimensional imaging (TDI) system commonly used to evaluate anatomical parameters of breast form and volume. This study uniquely employs TDI to evaluate the position of breast landmarks over time to objectively assess ptosis following ADM and non- ADM-based breast reconstructions. The following breast landmarks will be identified using a Vectra algorithm and confirmed by a trained medical assistant: sternal notch (Sn), nipple (N), and inframammary fold (IMF). Breast ptosis, defined as depression of breast tissue with respect to the IMF, will be objectively assessed as the relative position of nipple to the inferior margin. Changes in Sn-IMF and N-IMF lengths will be normalized across implant size. This will provide an indication of the amount of breast ptosis experienced by ADM and non-ADM cohorts per unit volume of prosthesis.

SECONDARY OUTCOMES:
Infection | 90 days post-operatively.
  Surgical site infection as defined by criteria described by centers for disease control and prevention (CDC).
Self reported outcomes | Post-surgical, follow-up intervals extending to one year following reconstruction.
  Patient subjective evaluation of aesthetic outcome via Breast-Q questionnaire.

IPD SHARING:
Plan to Share IPD: No
No intention to share individual participant data to other researchers.